CLINICAL TRIAL: NCT06684743
Title: A Pragmatic Randomized Trial to Evaluate the Vaccine Effectiveness of Abrysvo® for Preventing RSV Hospitalizations in Adults Aged 18 Years or Above
Brief Title: Vaccine Effectiveness of a Bivalent RSV Prefusion F Protein-Based Vaccine for Preventing RSV Hospitalizations in Adults
Acronym: DAN-RSV
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAN-RSV; 2024-516600-42-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: RSV
Keywords: RSV; Vaccination; Pragmatic; Registry; Lower respiratory tract disease; Respiratory tract disease; Respiratory; Cardiovascular
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSV prefusion F protein-based vaccine (RSV vaccine) (Experimental): RSV vaccine single injection at day 0
  Interventions: Biological: RSV prefusion F protein-based vaccine
- No RSV vaccine (control) (No Intervention): Control arm, no RSV vaccine

INTERVENTIONS:
Biological: RSV prefusion F protein-based vaccine — For this arm, the RSV prefusion F protein-based vaccine Abrysvo® will be used
  Other Names: RSVpreF vaccine
  Arms: RSV prefusion F protein-based vaccine (RSV vaccine)

SUMMARY:
The purpose of this pragmatic randomized trial is to evaluate the vaccine effectiveness of bivalent RSV prefusion F vaccine (RSV vaccine) in adults. Participants will be randomized 1:1 to either RSV vaccine or no RSV vaccine.

DETAILED DESCRIPTION:
The study is a pragmatic, registry-based, open-label, individually randomized trial. Administrative health registries will be used for data collection including baseline information, follow-up data, and safety monitoring. The study aims to randomize a total of 690,000 participants. Participants will be individually randomized 1:1 to receive either a bivalent RSV prefusion F vaccine (RSV vaccine) or no RSV vaccine. The trial is designed to assess the vaccine effectiveness of the RSV vaccine vs. no RSV vaccine on RSV-related and all-cause cardio-respiratory outcomes.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years and above
* Informed consent form has been signed and dated

Exclusion Criteria:

* There are no specific exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 690000 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Hospitalization for RSV-related respiratory tract disease | ≥14 days after initially booked vaccination/ information visit date up to 8 months

SECONDARY OUTCOMES:
RSV-related respiratory tract disease hospitalization | ≥14 days after actual vaccination date/ booked information visit date up to 8 months
  Primary outcome evaluated among the as-treated study population with balanced follow up time between study arms
Hospitalization for RSV-related lower respiratory tract disease | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Hospitalization for RSV-related respiratory tract disease by age groups | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Stratified by age groups (18-59, 60-74 years and 75+ years)
Hospitalization for RSV-related respiratory tract disease in subsequent seasons | From September 1, 2025 up to 9 months (2025/2026 season) and September 1, 2026 up to 9 months (2026/2027 season)
  Subsequent seasons (2025/2026 and 2026/2027 RSV seasons)
RSV-related hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
All-cause respiratory tract disease hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
RSV-related cardio-respiratory hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
All-cause cardio-respiratory hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
All-cause lower respiratory tract disease hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
All-cause hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
All-cause mortality | ≥14 days after initially booked vaccination/ information visit date up to 8 months

OTHER OUTCOMES:
Hospitalization for RSV-related respiratory tract disease stratified by RSV type | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Stratification by RSV type (A or B)
Total length of hospital stays due to respiratory tract infection with RSV infection | ≥14 days after initially booked vaccination/ information visit date up to 8 months
RSV or pneumonia hospitalization [composite endpoint] | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Based only on ICD-10 codes
Pneumonia hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Any hospitalization with RSV infection | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Cardiovascular disease hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Hospitalization requiring mechanical ventilation | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Intensive care unit hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Myocardial infarction hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Heart failure hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Stroke hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Influenza hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
COVID-19 hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Hospitalization for pneumococcal disease | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Any infectious disease hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
MACE (composite endpoint) | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Non-fatal myocardial infarction, heart failure hospitalization, stroke, and cardiovascular death
Laboratory-confirmed RSV infection | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Laboratory-confirmed influenza infection | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Laboratory-confirmed pneumococcal infection | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Laboratory-confirmed COVID-19 infection | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Cardio-respiratory mortality | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Respiratory mortality | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Cardiovascular mortality | ≥14 days after initially booked vaccination/ information visit date up to 8 months
In-hospital mortality | ≥14 days after initially booked vaccination/ information visit date up to 8 months
30-day mortality following hospital discharge for primary endpoint | ≥14 days after initially booked vaccination/ information visit date up to 8 months
Hospitalization for RSV-related lower respiratory tract disease in subsequent 2025/2026 and 2026/2027 RSV seasons | From September 1, 2025 up to 9 months (2025/2026 season) and September 1, 2026 up to 9 months (2026/2027 season)
RSV-related respiratory tract disease hospitalization by chronic obstructive pulmonary disease status | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Primary endpoint in patients with chronic obstructive pulmonary disease
New-onset dementia | ≥14 days after initially booked vaccination/ information visit date up to 10 years
RSV-related respiratory tract disease hospitalization by immunocompromised status | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Stratified by immunocompromised status. Analysis will be carried out as outlined in C3761080, EU PASS register number EUPAS1000000480
RSV-related lower respiratory tract disease hospitalization by immunocompromised status | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Stratified by immunocompromised status. Analysis will be carried out as outlined in C3761080, EU PASS register number EUPAS1000000480
All-cause respiratory tract disease hospitalization by immunocompromised status | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Stratified by immunocompromised status. Analysis will be carried out as outlined in C3761080, EU PASS register number EUPAS1000000480
All-cause lower respiratory tract disease hospitalization by immunocompromised status | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Stratified by immunocompromised status. Analysis will be carried out as outlined in C3761080, EU PASS register number EUPAS1000000480
RSV-related respiratory tract disease hospitalization by severe immunocompromised status | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Stratified by severe immunocompromised status. Analysis will be carried out as outlined in C3761080, EU PASS register number EUPAS1000000480
All-cause respiratory tract disease hospitalization by severe immunocompromised status | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Stratified by severe immunocompromised status. Analysis will be carried out as outlined in C3761080, EU PASS register number EUPAS1000000480
Atrial fibrillation hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Analysis will be carried out as outlined in C3761080, EU PASS register number EUPAS1000000480
Hospitalization for any cardiac arrythmia | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Analysis will be carried out as outlined in C3761080, EU PASS register number EUPAS1000000480
Hospitalization for pericarditis | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Analysis will be carried out as outlined in C3761080, EU PASS register number EUPAS1000000480
Hospitalization for myocarditis | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Analysis will be carried out as outlined in C3761080, EU PASS register number EUPAS1000000480
Asthma exacerbation hospitalization | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Analysis will be carried out as outlined in C3761080, EU PASS register number EUPAS1000000480
RSV-related respiratory tract disease hospitalization by hepatic or renal impairment status | ≥14 days after initially booked vaccination/ information visit date up to 8 months
  Among those with hepatic or renal impairment at baseline. Analysis will be carried out as outlined in C3761080, EU PASS register number EUPAS1000000480

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, PhD, MSc, MPH, Study Chair — Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte
Locations (3):
- Denmark (2):
  - Center for Translational Cardiology and Pragmatic Randomized Trials Department of Cardiology Copenhagen University Hospital - Herlev and Gentofte, Copenhagen
  - Danske Lægers Vaccinations Service, Søborg
- General Public Health Directorate of Galician Health Service, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
In this trial, baseline and endpoint data will be collected from Danish administrative health registries, which are subject to Danish legislation and can only be made available to a third party under certain conditions. Please contact the sponsor-investigator in case of any inquiries.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Lassen MCH, Johansen ND, Christensen SH, Aliabadi N, Skaarup KG, Modin D, Claggett BL, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Lindholm MG, Jensen AMR, Dons M, Bernholm KF, Davidovski FS, Duus LS, Ottosen CI, Nielsen AB, Borchsenius JH, Espersen C, Kose G, Fussing FH, Kober L, Solomon SD, Jensen JUS, Martel CJ, Gessner BD, Schwarz C, Gonzalez E, Skovdal M, Moulton LH, Zhang P, Begier E, Biering-Sorensen T. RSV Prefusion F Vaccine for Prevention of Hospitalization in Older Adults. N Engl J Med. 2026 Jan 8;394(2):138-151. doi: 10.1056/NEJMoa2509810. Epub 2025 Aug 30. PMID 40888695
- [Derived] Lassen MCH, Johansen ND, Christensen SH, Aliabadi N, Skaarup KG, Modin D, Claggett BL, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Lindholm MG, Jensen AMR, Dons M, Bernholm KF, Davidovski FS, Duus LS, Ottosen CI, Nielsen AB, Borchsenius JH, Espersen C, Kose G, Fussing FH, Pareek M, Kober L, Solomon SD, Jensen JUS, Martel CJ, Gessner BD, Schwarz C, Gonzalez E, Skovdal M, Moulton LH, Zhang P, Begier E, Biering-Sorensen T. Bivalent RSV Prefusion F Protein-Based Vaccine for Preventing Cardiovascular Hospitalizations in Older Adults: A Prespecified Analysis of the DAN-RSV Trial. JAMA. 2025 Oct 28;334(16):1431-1441. doi: 10.1001/jama.2025.15405. PMID 40884493
- [Derived] Lassen MCH, Christensen SH, Johansen ND, Aliabadi N, Skaarup KG, Modin D, Claggett BL, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Lindholm MG, Kober L, Solomon SD, Staehr Jensen JU, Martel CJ, Schwarz C, Gonzalez E, Skovdal M, Moulton LH, Zhang P, Gessner BD, Begier E, Biering-Sorensen T. A pragmatic individually randomized trial to evaluate bivalent RSV prefusion F protein-based vaccine effectiveness for preventing RSV hospitalizations in adults aged 60 years or above (DAN-RSV): Rationale and trial design. Am Heart J. 2026 Jan;291:14-25. doi: 10.1016/j.ahj.2025.07.068. Epub 2025 Jul 28. PMID 40738309